CLINICAL TRIAL: NCT05107596
Title: Preliminary Evaluation of 64Cu-DOTA-ECL1i in Patients Post-ST-Elevation Myocardial Infarction(STEMI)
Brief Title: Evaluation of CCR2 in Patients Post Myocardial Infarction
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201807140
Record Dates: First submitted 2021-10-07; First posted 2021-11-04 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Post ST Elevation Myocardial Infarction/ Heart Attack (Active Comparator): Image patients who have had a heart attack
  Interventions: Drug: 64Cu-DOTA-ECL1i
- Sarcoidosis (Active Comparator): Image patients who have Sarcoidosis
  Interventions: Drug: 64Cu-DOTA-ECL1i
- Myocarditis (Active Comparator): Image patients with Myocarditis
  Interventions: Drug: 64Cu-DOTA-ECL1i
- Cardiomyopathy (Active Comparator): Image patients with cardiomyopathy
  Interventions: Drug: 64Cu-DOTA-ECL1i
- Infected Cardiovascular Implantable Electronic Devices (Active Comparator): Image patients with cardiovascular implanted medical devices
  Interventions: Drug: 64Cu-DOTA-ECL1i
- Healthy Volunteers (Active Comparator): Image healthy volunteers
  Interventions: Drug: 64Cu-DOTA-ECL1i

INTERVENTIONS:
Drug: 64Cu-DOTA-ECL1i — Inject PET Radioisotope for imaging
  Other Names: Imaging drug

SUMMARY:
To determine the feasibility of 64Cu-DOTA-ECL1i, an investigational PET imaging drug, at the cellular level in the myocardium for individuals who have suffered a heart attack or who have other inflammatory heart disease.

DETAILED DESCRIPTION:
To determine the feasibility of 64Cu-DOTA-ECL1i to detect CCR2+monocytes and macrophages which are cells that are responsible for protecting tissues from foreign substances in the myocardium by PET/MR and PET/CT.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Volunteers:
2. Age 21 to 80 years of either sex, any race
3. Capable of lying still and supine within the PET/CT and PET/MR scanner for 1 hour and follow instructions for breathing protocol during the CT portion
4. No illicit drug use or other inhaled drug use (including pharmacologic agents, recreational agents, or illicit drugs) within the past year
5. No known history of cardiac. pulmonary, hepatic, or renal disease or diabetes
6. No history of claustrophobia or other preventing condition that has previously or would interfere with completion of protocol-specified imaging sessions
7. Able to comprehend and willing to follow instructions for the study procedures as called for by the protocol.

Inflammatory Heart Disease

1. Age 21 to 80 years of either sex, any race who have suffered a STEMI within the past 6 months as well as other forms of inflammatory heart disease including sarcoidosis, myocarditis, cardiomyopathy, injected cardiovascular implantable electronic devices pacemakers/LVAD
2. Are clinically stable to undergo imaging with either PET/MR or PET/CT.
3. Capacity to give written informed consent and ability to follow study procedures
4. Pre-menopausal women must have a negative urine pregnancy test within 24 hours prior to the administration of 64-Cu-DOTA-ECL1i.

Exclusion Criteria:

Healthy volunteers:

1. Currently enrolled in another study using an investigational drug
2. Angina
3. Uncontrolled heart failure
4. uncontrolled hypertension baseline hypotension below 90/50
5. Has any condition that in the opinion of the PI or designee that could increase risk to the subject
6. Is deemed likely to be unable to perform all research procedures
7. Have contraindications to PET/CT imaging like claustrophobia
8. Have contraindication to gadolinium
9. Pregnant or breastfeeding
10. Currently using recreational drubs
11. Body weight of more than 300 lbs
12. Active symptoms or history of cardiac, pulmonary, hepatic or renal disease or diabetes
13. currently taking any prescription medications
14. Presence of an implanted device incompatible with CT or MRI scanning Inflammatory Heart Disease

1) Clinically unstable including post MI angina, uncontrolled heart failure, sever hypertension, hypotension AV block 2) Has any condition that in the opinion of the PI could increase risk to the subject 3) Claustrophobia 4) contraindication to gadolinium contrast 5) Pregnant 6) Currently using recreational drugs 7) Body Weight more than 300 lbs 8) Currently enrolled in another study

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-11-24 (Actual); Primary Completion 2025-11-24 (Estimated); Study Completion 2025-11-24 (Estimated)

PRIMARY OUTCOMES:
Number of participants who have heart disease as shown in the images | 1 or 2 days
  PET images will be reconstruction using an iterative algorithm that incorporates resolution recovery, and will be corrected for attenuation using their respective CT or MR data sets

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States